CLINICAL TRIAL: NCT06630884
Title: Inflammatory Challenge and Fear Extinction: A Model to Enhance Understanding of Posttraumatic Stress Disorder
Brief Title: Inflammatory Challenge and Fear
Acronym: LIFE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Northern California Institute of Research and Education (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R01MH135076 (NIH); R01MH135076 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; posttraumatic stress; inflammation; fear
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Inflammation | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Polysaccharide typhoid vaccine (Experimental): Participants in this condition will receive an injection of 0.5ml Salmonella typhi capsular polysaccharide vaccine (Sanofi Pasteur, SA), which contains 25μg of purified Vi polysaccharide in a colorless isotonic phosphate buffered saline (pH 7±0.3), 4.150mg of sodium chloride, 0.065mg of disodium phosphate, 0.023mg of monosodium phosphate and 0.5ml of sterile water for injection.
  Interventions: Biological: Typhoid VI Polysaccharide Vaccine Injectable Solution
- Saline Placebo Arm (Placebo Comparator): Participants in this condition will receive and injection of 0.5ml of saline.
  Interventions: Other: Saline Placebo (0.5mL injection)

INTERVENTIONS:
Biological: Typhoid VI Polysaccharide Vaccine Injectable Solution — Salmonella typhi capsular polysaccharide vaccine (Typhoid Vi Polysaccharide Vaccine): Each dose of 0.5ml Salmonella typhi capsular polysaccharide vaccine (Sanofi Pasteur, SA) is formulated to contain 25μg of purified Vi polysaccharide in a colorless isotonic phosphate buffered saline (pH 7±0.3), 4.150mg of sodium chloride, 0.065mg of disodium phosphate, 0.023mg of monosodium phosphate and 0.5ml of sterile water for injection. It is indicated for use by humans aged 2 years and older for protection against typhoid fever.
  Arms: Polysaccharide typhoid vaccine
Other: Saline Placebo (0.5mL injection) — The placebo injection will consist of 0.5mL of saline.
  Arms: Saline Placebo Arm

SUMMARY:
The goal of this study is to learn if short-term changes in the immune system alter how we process information and experience fear. The main questions it aims to answer are:

Do people who receive typhoid vaccine respond differently than those who receive a placebo saline vaccine? Do people who receive typhoid vaccine experience changes in how they think and feel?

Participants will:

Attend four appointments at the San Francisco VA Health Care System;

Receive typhoid vaccine or placebo at one of the visits;

Have their physiological responding measured while listening to sounds;

Complete questionnaires and psychological tests.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a chronic disorder affecting more than 8% of the general population and two-three times as many women as men. Deficits in fear responding play a critical role in PTSD. Interventions that target fear responding are first-line treatments for PTSD, but they are only partially effective. To develop new and enhanced interventions, we need a better understanding of the factors that influence fear responding in PTSD in both females and males. One such factor is inflammation, which is elevated in response to acute psychological stress and in PTSD. Preclinical models indicate that elevated inflammation in general, and elevated levels of the pro-inflammatory cytokine interleukin-6 (IL-6) in particular, can impair fear responses. People with PTSD and women may be more sensitive to the effects of inflammatory activity on fear responses. The long-term goal is to uncover the mechanistic role that inflammation plays in PTSD in order to identify effective primary and adjunctive anti-inflammatory interventions. The objective in this proposal is to determine the effects of acute inflammatory challenge on fear responding in trauma-exposed women and men with and without PTSD. The central hypothesis is that acute inflammatory challenge will alter fear responding, with particularly strong effects in people with chronic PTSD and women. The aims are to: 1) determine the effects of acute inflammatory challenge on fear responding in individuals with and without PTSD; 2) examine if increases in inflammatory activity mediate associations between acute inflammatory challenge and fear responses; and 3) elucidate sex differences in the effects of acute inflammatory challenge on fear responses. In the proposed study, we will use polysaccharide typhoid vaccine, which preliminary data support as a robust acute inflammatory challenge, and a fear learning paradigm that we have used in >200 people with PTSD. Participants will first undergo physiological testing of fear responses. Then, three days later, participants will receive either vaccine or placebo and undergo more tests, including physiological tests. One week later, we will test physiological responses again. Inflammatory markers will be measured at baseline, twice on the the vaccine/placebo day, and once at the one-week follow-up visit. This proposal is significant and innovative because it would be the first study to examine the effects of acute inflammatory activity on fear responses in trauma-exposed individuals with and without PTSD, and it has potential to elucidate biological mechanisms of impaired fear responses, uncover sex differences, and point us in the direction of novel interventions to treat PTSD.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

1. Aged 18-60 years old
2. Trauma Exposed
3. Current PTSD/No history of PTSD

Exclusion Criteria:

1. Contraindications to typhoid vaccine
2. Conditions associated with inflammation
3. Pregnancy or plans to become pregnant in next three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Skin conductance response (SCR) | SCR will be assessed at baseline, 4.5 hours, and one week after vaccine/placebo.
  Skin conductance level (SCL)will be sampled at 1000 Hz beginning 2 s prior to the conditioned stimulus (CS) onset and continuing until 6 s following CS offset. The skin conductance response (SCR) score for each CS interval will be obtained by subtracting the mean SCL for the 2 s preceding CS onset from the peak during the 8 s CS interval.

SECONDARY OUTCOMES:
Heart rate | HR will be assessed at baseline, 4.5 hours, and one week after vaccine/placebo.
  HR will be calculated by subtracting average HR of every 0.5 s interval during 6 s before CS (baseline) from peak HR during 0.5 s interval of 8 s after CS onset (response).
Eyeblink electromyography (EMG) | Eyeblink EMG will be assessed at baseline, 4.5 hours, and one week after vaccine/placebo.
  EMG will be calculated by subtracting the mean signal amplitude during 2 s preceding CS onset (baseline) from the peak during the 8 s CS interval (response).

CONTACTS AND LOCATIONS:
Overall Officials: Aoife O'Donovan, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical, biological, and psychophysiological data will be acquired from 120 individuals with PTSD and 120 individuals without PTSD. Demographic data will be self-reported. Clinical data will include information from validated semi-structured clinical interviews and validated self-report measures assessing symptoms of PTSD and other psychiatric disorders. Biological data will include levels of eleven inflammatory markers derived from five blood draws for each participant. Psychophysiological data will include skin conductance level, heart rate (HR), and HR variability (HRV) assessed 34 times for each participant.
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: Related Info — http://odonovanlab.ucsf.edu